CLINICAL TRIAL: NCT07070752
Title: Multicenter, Open-Label, Randomized, Controlled Study of Non-Inferior Immunogenicity of GP40321 (Solution for Subcutaneous Injection, 100 U/mL; GEROPHARM LLC, Russia) and Apidra® SoloStar® (Solution for Subcutaneous Injection, 100 U/mL; Sanofi-Aventis Deutschland GmbH, Germany) in Type 1 Diabetes Mellitus Patients
Brief Title: Evaluation of Insulin Glulisine (GP40321) Compared to Insulin Glulisine (Apidra® SoloStar®) in Type 1 Diabetes Mellitus Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Geropharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GP40321-P4-03-01
Record Dates: First submitted 2025-07-09; First posted 2025-07-17 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Type 1 Diabetes Mellitis
MeSH Terms: interventions — insulin glulisine; Insulin Glargine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GP40321 (Experimental)
  Interventions: Drug: GP40321; Drug: RinGlar®
- Apidra® SoloStar® (Active Comparator)
  Interventions: Drug: Apidra® SoloStar®; Drug: RinGlar®

INTERVENTIONS:
Drug: GP40321 — GP40321, solution for subcutaneous injection, 100 U/mL (GEROPHARM LLC, Russia)
  Other Names: insulin glulisine
  Arms: GP40321
Drug: Apidra® SoloStar® — Apidra® SoloStar®, solution for subcutaneous injection, 100 U/mL (Sanofi-Aventis Deutschland GmbH, Germany)
  Other Names: insulin glulisine
  Arms: Apidra® SoloStar®
Drug: RinGlar® — Patients also receive long-acting basal insulin therapy (insulin glargine 100 U/mL) throughout the study
  Other Names: insulin glargine

SUMMARY:
The goal of this clinical trial is to demonstrate the non-inferior immunogenicity of GP40321 compared to Apidra® SoloStar® at a concentration of 100 U/mL in type 1 diabetes mellitus patients. The main questions it aims to answer are:

* What is the immunogenicity of GP40321 and Apidra® SoloStar®?
* What are the efficacy and safety of GP40321 and Apidra® SoloStar®?

Researchers will compare the immunogenicity, efficacy and safety parameters of GP40321 and Apidra® SoloStar®.

Participants will:

• Visit the clinic 9 times: once for screening, 3 times during dose titration (plus 2 telephone contacts) and 5 times during the stable dose treatment period.

ELIGIBILITY:
Inclusion Criteria

* Signed informed consent to participate in the study.
* Male or female sex.
* Age ≥18 years at the time of providing informed consent.
* Diagnosis of type 1 diabetes mellitus (T1DM) for ≥12 months prior to the Screening Visit.
* Body Mass Index (BMI) between 18.5-35.0 kg/m² at the Screening Visit.
* Stable basal-bolus insulin therapy for ≥6 months prior to the Screening Visit, including:

  1. Insulin glargine (100 U/mL)

     IN COMBINATION WITH
  2. Insulin aspart (100 U/mL) OR
  3. Insulin lispro (100 U/mL) OR
  4. Insulin glulisine (100 U/mL)
* HbA1c level ≥6.5% and ≤10%, measured at screening.
* Willingness and ability to comply with study procedures, including the 7-point glycemic profile and self-monitoring of blood glucose, as well as protocol-specified restrictions and prohibitions.

Exclusion Criteria

Related to Insulin Therapy

* Contraindications to insulin glulisine or insulin glargine therapy.
* History of hypersensitivity to any component of the investigational product or significant allergic reactions to medications, including any type of insulin.
* Severe insulin resistance (defined as insulin requirement >1.5 U/kg/day).
* Change of the INN (International Nonproprietary Name) of bolus or basal insulin within 6 months prior to Screening.
* Use of biosimilar insulin products within 6 months prior to Screening, except for those from GEROPHARM LLC.
* Use of insulin pump therapy within 6 months prior to Screening or planned initiation during the study.
* Use of systemic glucocorticoids at supraphysiologic doses for ≥7 days within 3 months prior to Screening.
* Use of hypoglycemic drugs other than insulin products, including injectable glucagon-like peptide-1 receptor agonists (aGLP-1), within 3 months prior to Screening or planned initiation during the study.

Related to T1DM progression and subject health risk

* History of or screening-identified chronic T1DM complications, including:

  1. Proliferative diabetic retinopathy, which may require intervention during the study period (laser ablation, surgical treatment, injectable drugs, etc.), in the opinion of the Investigator;
  2. Severe diabetic peripheral or autonomic neuropathy, in the opinion of the Investigator;
  3. Chronic kidney disease (including diabetic nephropathy) with an estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m²;
  4. Current diabetic foot syndrome that may require intervention during the study period (surgical treatment, wound rehabilitation, limb relief, adjuvant therapy, antibacterial therapy, etc.).
* Acute T1DM complications within 3 months prior to Screening or identified during screening, including:

  1. Episode of severe hypoglycemia (which required the help of another person or hospitalization);
  2. Episode of diabetic ketoacidosis;
  3. Episode of hyperosmolar hyperglycemic state.
* More than 15 episodes of mild hypoglycemia (symptomatic or asymptomatic) within 1 month prior to Screening or identified during screening.

Related to comorbidities and subject health risk

* Conditions affecting hemoglobin level assessment (e.g., history of hemoglobinopathy or hemolytic anemia, blood transfusion within 3 months prior to Screening); anemia that cannot be corrected before subject enrollment.
* Significant blood loss within 3 months prior to Screening, including but not limited to:

  1. Blood donation;
  2. Extensive surgery or trauma resulting in significant blood loss.
* Abnormal results of the following screening laboratory tests:

  1. hemoglobin level <9.0 g/dL (SI system: <90 g/L);
  2. hematocrit <30%;
  3. ALT or AST >2 upper limits of normal (ULN) or either ALT or AST >3× ULN;
  4. serum bilirubin level >2 ULN (excluding subjects with previously diagnosed Gilbert's syndrome).
* History of or clinically significant condition identified during screening, including but not limited to:

  1. Unstable angina, myocardial infarction, arrhythmia requiring medical treatment, or congestive heart failure class III or IV according to the New York Heart Association (NYHA) classification within 1 year prior to the Screening Visit;
  2. Stroke or transient ischemic attack within 6 months prior to the Screening Visit.
* Pregnancy or breastfeeding.

Related to immunogenicity assessment

* Regular use of immunotropic therapy or any other medications that may affect the patient's immune status.
* Vaccination within 3 months prior to the anticipated randomization date or planned during the study period.
* History of autoimmune diseases other than vitiligo and controlled autoimmune diseases that are part of autoimmune polyglandular syndrome (types 1-3), with the exception of adrenal insufficiency.
* A burdened allergic history, which, according to the Investigator, may affect the results of the study or endanger the patient's safety.
* Full recovery from an acute inflammatory illness less than 4 weeks before the Screening Visit.
* Incomplete recovery from surgery or surgical intervention planned for the period of the patient's participation in the study.
* Positive serological test results for infections:

  1. Human immunodeficiency virus (HIV-1/2 antibodies);
  2. Hepatitis B (surface antigen);
  3. Hepatitis C (antibodies to hepatitis C virus antigens).
* History or presence of oncological and/or oncohematological diseases not in full 5-year remission at the Screening Visit.
* History of organ and/or bone marrow transplantation (except for corneal transplantation performed ≥3 months prior to Screening).

Related to risk of protocol non-compliance

* Planned hospitalization for any reason during the study period.
* Mental, physical, or other conditions that prevent the subject from adequately assessing their behavior or properly complying with the study protocol, including a history of mental illness.
* Current or past (within three years prior to the first administration of the investigational product) history of alcohol, drug, medication, and/or substance abuse.
* Participation in another clinical study within 28 days prior to Screening or planned participation during the current study.
* Any other conditions that, in the opinion of the Investigator, represent a contraindication for study participation (i.e., may adversely affect the subject's condition if they participate, may interfere with study procedures, or affect the interpretation of study results). In case of doubt, the Investigator should consult the Medical Expert for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2023-04-14 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2023-11-28 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who develop an immune response | From screening to the end of treatment at Week 26
  The proportion of patients who develop an immune response during the study.

SECONDARY OUTCOMES:
Change in mean anti-insulin antibodies (AIA) level | From screening to the end of treatment at Week 26
  Change in mean anti-insulin antibodies (AIA) level after 26 weeks compared with baseline at Screening.
Change in mean neutralizing anti-insulin antibodies (nAIA) level | From screening to the end of treatment at Week 26
  Change in mean neutralizing anti-insulin antibodies (nAIA) level after 26 weeks compared with baseline at Screening.
Incidence of nAIA in nAIA-naïve subjects | From screening to the end of treatment at Week 26
  Incidence of nAIA during 26 weeks of insulin therapy in nAIA-naïve subjects.
Proportion of patients with clinically significant immune response | From screening to the end of treatment at Week 26
  Proportion of patients who develop a clinically significant immune response within 26 weeks.
Change in mean HbA1c level | From screening to the end of treatment at Week 26
  Change in mean HbA1c level after 26 weeks compared with baseline at Screening.
Proportion of patients with HbA1c ≤7.0% | From screening to the end of treatment at Week 26
  Proportion of patients with HbA1c ≤7.0% in the absence of nocturnal and severe hypoglycemia after 26 weeks.
Proportion of patients with reached individual target HbA1c | From screening to the end of treatment at Week 26
  Proportion of patients who reach their individual target HbA1c after 26 weeks.
Change in mean fasting plasma glucose (FPG) | From screening to the end of treatment at Week 26
  Change in mean fasting plasma glucose (FPG) after 26 weeks compared with baseline at Screening.
Change in mean values of the 7-point glycemic profile | From screening to the end of treatment at Week 26
  Change in mean values of the 7-point glycemic profile after 22 weeks of stable-dose insulin therapy compared with baseline at Screening.
Change in mean values of the 7-point glycemic profile | From the end of the dose titration period to the end of treatment at Week 26
  Change in mean values of the 7-point glycemic profile after 22 weeks of stable-dose insulin therapy compared with the end of the titration period.
Change in mean total daily insulin dose | From the end of the dose titration period to the end of treatment at Week 26
  Change in mean total daily insulin dose after 22 weeks of stable-dose insulin therapy compared with the end of the titration period.
Change in mean body weight | From screening to the end of treatment at Week 26
  Change in mean body weight at Week 26 compared with baseline at Screening.
Treatment satisfaction | From screening to the end of treatment at Week 26
  Assessment of satisfaction with diabetes mellitus treatment using the DTSQs questionnaire after 26 weeks.
Assessment of safety | From screening to the end of treatment at Week 26
  - Frequency and severity of adverse events (AE)/serious adverse events (SAE) based on abnormalities in vital signs, ECG readings, and laboratory tests. -Separate assessment of the following AE/SAE: a. the frequency of hypoglycemia; b. the frequency of ketoacidosis; c. the frequency of injection site reactions; d. the frequency of allergic reactions. - Changes in vital signs compared to baseline. - Changes in laboratory test results compared to baseline.

CONTACTS AND LOCATIONS:
Locations (16):
- Russia (16):
  - RZD-Medicine Clinical Hospital of Chelyabinsk, Chelyabinsk
  - Interregional Clinical and Diagnostic Center, Kazan'
  - Krasnoyarsk State Medical University named after Professor V.F. Voino-Yasenetsky, Ministry of Health of the Russian Federation, Krasnoyarsk
  - National Medical Research Center of Endocrinology of the Ministry of Health of the Russian Federation, Moscow
  - "Endocrinological Dispensary of the Moscow City Health Department", Moscow
  - Almazov National Medical Research Center of the Ministry of Health of the Russian Federation, Saint Petersburg
  - X7 Research, LLC, Saint Petersburg
  - City Multidisciplinary Hospital No. 2, Saint Petersburg
  - "City polyclinic No. 117", Saint Petersburg
  - St. Elizabeth City Hospital of the Holy Martyr, Saint Petersburg
  - "City polyclinic No. 112", Saint Petersburg
  - "Eco-Safety" Research Center, LLC, Saint Petersburg
  - City Pokrovskaya Hospital, Saint Petersburg
  - "City polyclinic No. 4", Saint Petersburg
  - "Diabetes Center", LLC, Samara
  - Volgograd Regional Clinical Hospital No. 1, Volgograd

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Drai R, Galstyan G, Karonova T, Protsenko E, Parfenova T, Arefeva A, Matvienko I, Iliushchenko D, Makarenko I. Immunogenicity, efficacy and safety of a biosimilar insulin glulisine compared with originator in adults with type 1 diabetes mellitus: A phase III randomised clinical trial. Diabetes Obes Metab. 2026 Mar;28(3):1791-1799. doi: 10.1111/dom.70360. Epub 2025 Dec 9. PMID 41366610